CLINICAL TRIAL: NCT04242199
Title: A Phase 1 Study Exploring the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of INCB099280 in Participants With Select Advanced Solid Tumors
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of INCB099280 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 99280-112; 2019-004967-35 (EudraCT Number)
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor; MSI-H/dMMR Tumors; Cutaneous Squamous Cell Carcinoma; Urothelial Carcinoma; Cervical Cancer; HepatoCellular Carcinoma; Esophageal Squamous Cell Carcinoma; Merkel Cell Carcinoma; Small-cell Lung Cancer; Mesothelioma; PD-L1 Amplified Tumor (9p24.1); Nasopharyngeal Carcinoma
Keywords: Advanced Solid Tumor
MeSH Terms: conditions — Carcinoma, Transitional Cell; Uterine Cervical Neoplasms; Carcinoma, Hepatocellular; Esophageal Squamous Cell Carcinoma; Carcinoma, Merkel Cell; Small Cell Lung Carcinoma; Mesothelioma; Nasopharyngeal Carcinoma

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts. Part 1 is a dose-escalation design to identify the maximum tolerant dose and/or pharmacologically active dose for INCB099280. Part 2 is an expansion at 1 or more dose levels to further explore safety, preliminary efficacy, pharmacokinetic, and pharmacodynamic effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants with select solid tumors who are immunotherapy treatment-naive
  Interventions: Drug: INCB099280
- Cohort 2 (Experimental): Participants with high microsatellite instability (MSI-H) or deficient mismatch repair (dMMR) tumors who are immunotherapy treatment-naïve.
  Interventions: Drug: INCB099280
- Cohort 3 (Experimental): Participants with progression of any solid tumor treated with an approved anti-PD-1 monoclonal antibody therapy
  Interventions: Drug: INCB099280

INTERVENTIONS:
Drug: INCB099280 — INCB099280 administered orally in 25 mg or 100 mg tablets once daily or twice daily on each day of each 28-day cycle

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics, pharmacodynamics, and early clinical activity of INCB099280 in participants with select solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Must have disease progression after treatment with available therapies that are known to confer clinical benefit or must be intolerant to or ineligible for standard treatment.
* Histologically confirmed advanced solid tumors (protocol-defined select solid tumors) with measurable lesions per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) that are considered nonamenable to surgery or other curative treatments or procedures.
* Eastern Cooperative Oncology Group performance status score of 0 or 1.
* Life expectancy > 12 weeks.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Laboratory values outside the Protocol-defined ranges.
* Clinically significant cardiac disease.
* History or presence of an electrocardiogram that, in the investigator's opinion, is clinically meaningful.
* Untreated brain or central nervous system (CNS) metastases or brain or CNS metastases that have progressed (eg, evidence of new or enlarging brain metastasis or new neurological symptoms attributable to brain or CNS metastases).
* Known additional malignancy that is progressing or requires active treatment.
* Has not recovered to ≤ Grade 1 or baseline from toxic effects of prior therapy (including prior IO) and/or complications from prior surgical intervention before starting study treatment.
* Prior receipt of an anti-PD-L1 therapy.
* Treatment with anticancer medications or investigational drugs within protocol-defined intervals before the first administration of study drug.
* A 28-day washout for systemic antibiotics is required.
* Probiotic usage while on study and during screening is prohibited.
* Active infection requiring systemic therapy.
* Known history of Human Immunodeficiency Virus (HIV)
* Evidence of hepatitis B virus or hepatitis C virus infection or risk of reactivation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Up to approximately 25 months
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug up to 30 days after last dose of study drug.

SECONDARY OUTCOMES:
Cmax of INCB099280 | Up to approximately 3 months
  Maximum observed plasma concentration
tmax of INCB099280 | Up to approximately 3 months
  Time to maximum plasma concentration
Cmin of INCB099280 | Up to approximately 3 months
  Minimum observed plasma concentration over the dose interval
AUC0-t of INCB099280 | Up to approximately 3 months
  Area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t
t½ of INCB099280 | Up to approximately 3 months
  Apparent terminal-phase disposition half-life
λz of INCB099280 | Up to approximately 3 months
  Terminal elimination rate constant
CL/F of INCB099280 | Up to approximately 3 months
  Oral dose clearance
Vz/F of INCB099280 | Up to approximately 3 months
  Apparent oral dose volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (21):
- United States (5):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Upmc Cancercenter, Pittsburgh, Pennsylvania
  - Md Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- Australia (4):
  - Chris Obrien Lifehouse, Camperdown, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - Nucleus Network Pty Ltd, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Belgium (5):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Institut Jules Bordet Clinical Trials Conduct Unit, Brussels
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Ghent University Hospital, Ghent
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
- France (5):
  - Institut de Cancerologie de L Ouest - Site Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Chu Hopital de La Timone, Marseille
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy, Villejuif
- Japan (2):
  - National Cancer Center Hospital East, Chiba
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data